CLINICAL TRIAL: NCT01953926
Title: An Open-Label, Phase 2 Basket Study of Neratinib in Patients With Solid Tumors With Somatic Activating HER Mutations
Brief Title: Basket Study of Neratinib in Participants With Solid Tumors Harboring Somatic HER2 or EGFR Exon 18 Mutations
Acronym: SUMMIT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated to align with the sponsor's current development plans for neratinib. The decision was not based on any new efficacy or safety data for neratinib.
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMA-NER-5201; 2013-002872-42 (EudraCT Number)
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Solid Tumors Harboring Somatic HER2 or EGFR Exon 18 Mutations
Keywords: Neratinib; Nerlynx; Breast; Solid Tumors; Cancer; HER2 mutations; EGFR mutations; Fulvestrant; Trastuzumab; Cervical; Salivary; ERBB2; Exon 18; Metastatic; HR Positive; Lung; Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung | interventions — neratinib; Fulvestrant; Trastuzumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Neratinib monotherapy (Experimental): Neratinib monotherapy in HER2 mutated cancers including cervical, salivary gland, and lung cancers containing EGFR exon 18 mutations.
  Cohorts closed to enrollment in prior amendments: HER2 mutant cancers including bladder/urinary, colorectal, endometrial, breast HR-positive, TNBC HR-negative, lung, gastroesophageal, biliary, and ovarian; HER3 mutant solid tumor NOS; HER4 mutant solid tumor NOS; fibrolamellar carcinoma and EGFR brain.
  Interventions: Drug: Neratinib
- Neratinib and Trastuzumab (Experimental): Neratinib and Trastuzumab in HER2 mutated (TNBC, HR-negative) breast cancers.
  Cohorts closed to enrollment in in prior amendments: colorectal, lung cancer HER2 mutant.
  Interventions: Drug: Neratinib; Drug: Trastuzumab
- Neratinib, Fulvestrant and Trastuzumab (Randomized) (Experimental): Neratinib, Fulvestrant and Trastuzumab or Fulvestrant and Trastuzumab or Fulvestrant alone in HER2 mutated (HR-positive with prior CDK4/6i) breast cancers.
  Interventions: Drug: Neratinib; Drug: Fulvestrant; Drug: Trastuzumab
- Neratinib, Fulvestrant and Trastuzumab (Non-Randomized) (Experimental): Neratinib, Fulvestrant and Trastuzumab in HER2 mutated (HR-positive with or without CDK4/6i) breast cancers.
  Interventions: Drug: Neratinib; Drug: Fulvestrant; Drug: Trastuzumab
- Neratinib and Paclitaxel (Experimental): Neratinib and Paclitaxel in HER2 mutated bladder/urinary tract cancers.
  Interventions: Drug: Neratinib; Drug: Paclitaxel
- Neratinib and Fulvestrant (Experimental): Neratinib and Fulvestrant in HER2 mutated (HR-positive) breast cancers.
  Interventions: Drug: Neratinib; Drug: Fulvestrant

INTERVENTIONS:
Drug: Neratinib — 240 mg administered orally, once daily with food, continuously in 28 day cycles
  Other Names: Nerlynx
Drug: Fulvestrant — 500 mg administered as two 5 mL injections on Days 1, 15, and 29; then once every 4 weeks thereafter month, then Day 1 of every 4 week cycle
  Other Names: Faslodex
  Arms: Neratinib and Fulvestrant; Neratinib, Fulvestrant and Trastuzumab (Non-Randomized); Neratinib, Fulvestrant and Trastuzumab (Randomized)
Drug: Trastuzumab — Initial dose of 8 mg/kg of trastuzumab administered IV on Day 1, followed by 6 mg/kg IV once every 3 weeks thereafter
  Other Names: Herceptin
  Arms: Neratinib and Trastuzumab; Neratinib, Fulvestrant and Trastuzumab (Non-Randomized); Neratinib, Fulvestrant and Trastuzumab (Randomized)
Drug: Paclitaxel — 80mg/m^2 administered IV on Days 1, 8, and 15 of every 4 week cycle
  Other Names: Taxol
  Arms: Neratinib and Paclitaxel

SUMMARY:
This is an open-label, multicenter, multinational, Phase 2 basket study exploring the efficacy and safety of neratinib as monotherapy or in combination with other therapies in participants with HER (EGFR, HER2) mutation-positive solid tumors.

DETAILED DESCRIPTION:
This is an open-label, multicenter, multinational, Phase 2 basket study exploring the efficacy and safety of neratinib as monotherapy or in combination with other therapies in participants with HER (EGFR, HER2) mutation-positive solid tumors. The study has a basket design and includes several cohorts, either defined by an actionable somatic mutation or by actionable mutation and tumor histology, including HER2 mutant breast, HER2 mutant cervical, HER2 mutant salivary gland, and EGFR Exon 18 mutant Non-small cell lung cancers.

The trial will consist of a screening period, a treatment period, and an end of treatment visit occurring when neratinib is discontinued for any reason, a safety follow-up visit occurring 28 days after the last dose of neratinib and a survival follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Histologically confirmed cancers for which no curative therapy exists
* Documented HER2 or EGFR exon 18 mutation
* Participants must agree and commit to use appropriate methods of contraception as outlined in the protocol
* At least one measurable lesion, defined by RECIST v1.1

Exclusion Criteria:

* Participants harboring ineligible somatic HER2 mutations
* Prior treatment with any HER2-directed tyrosine kinase inhibitor (e.g., lapatinib, afatinib, dacomitinib, neratinib) is excluded with the following exception: patients with EGFR exon 18 mutated NSCLC who may have received afatinib, osimertinib, or other pan HER or EGFR TKIs remain eligible
* Participants who are receiving any other anticancer agents
* Symptomatic or unstable brain metastases
* Women who are pregnant or breast-feeding

There are additional inclusion and exclusion criteria. The study center will determine if criteria for participation are met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 582 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2023-01-02 (Actual); Study Completion 2023-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Scientific Officer, Study Director — Puma Biotechnology, Inc.
Locations (60):
- United States (30):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - City of Hope, Duarte, California
  - University of California, San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Stanford Cancer Center, Palo Alto, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Kaiser Permanente NoCal (STRATA), Vallejo, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Washington University, St Louis, Missouri
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - UPMC Magee-Woman's Hospital, Women's Cancer Center, Pittsburgh, Pennsylvania
  - Saint Francis Cancer Center-Bon Secours, Greenville, South Carolina
  - The West Clinic, Germantown, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Gundersen Center for Cancer and Blood Disorders, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- Peter MacCallum Cancer Centre, East Melbourne, Victoria, Australia
- UZ Leuven, Leuven, Belgium
- British Columbia Cancer Center, Vancouver, British Columbia, Canada
- University Hospital, Rigshospitalet, Copenhagen, Denmark
- France (4):
  - Institut Gustave Roussy, Villejuif, Paris
  - Institut Bergonié, Bordeaux
  - Centre Leon Berard, Lyon
  - Institut Curie - Hopital Rene Huguenin, Saint-Cloud, Île-de-France Region
- St. Vincent's University Hospital, Dublin, Leinster, Ireland
- Israel (5):
  - Hadassah Medical Center, Jerusalem
  - Davidoff Cancer Center, Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Sourasky Medical Center, Tel Aviv
- Italy (4):
  - Azienda Socio Sanitaria Territoriale di Cremona, Cremona
  - Istituto Europeo di Oncologia (IEO) I.R.C.C.S., Milan
  - Fondazione Policlinico Universitario Gemelli I.R.C.C.S., Roma
  - AOU Citta della Salute e della Scienza di Torino, Torino
- Institute for Oncology and Radiology of Serbia, Belgrade, Serbia
- Yonsei University Health System, Serverance Hospital, Seodaemun-Gu, Seoul, South Korea
- Spain (9):
  - Hospital Universitario Quiron Dexeus, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitari Clinic Barcelona, Barcelona
  - Hospital Clinico Universitario San Carlos, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Madrid Sanchinarro (START Madrid), Madrid
  - Hospital Universitario Quiron Madrid, Madrid
  - Instituto Valenciano de Oncologia, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Puma Biotechnology is committed to sharing clinical trial data and information to help physicians and patients make informed treatment decisions, and to help qualified researchers advance scientific knowledge.
  In accordance with legal and regulatory requirements, Puma publishes study protocol information and clinical study results on clinical trial registries, including ClinicalTrials.gov and EU Clinical Trials Register. Puma also publishes information about clinical studies in peer-reviewed scientific journals and shares data in scientific meetings.
  Puma commits to safeguarding confidentiality and patient privacy throughout the clinical trial data and information sharing process. Any patient-level data will be anonymized to protect personally identifiable information.
  Qualified researchers and study participants may submit requests for other study documentation and clinical trial data to clinicaltrials@pumabiotechnology.com for consideration.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Clinical study documents and clinical trial data may be requested by qualified researchers and study participants for studies that have been completed for at least 18 months, and for which the indication of the drug has been approved in the US and/or EU, as applicable. Requests will be accepted for up to 24 months after the criteria described in this section are met.
Access Criteria: Requestors must provide organizational contact information; a detailed research plan, including outcomes; timeline for completion of the research; qualifications of the research team; funding source; and potential conflicts of interest.
  Puma will not provide access to patient-level data if there is a reasonable likelihood that individual patients could be identified, or in cases where confidentiality or consent provisions prohibit transfer of data or information to third parties. Additionally, Puma will not disclose information that jeopardizes intellectual property rights or divulges confidential commercial information.
URL: https://pumabiotechnology.com/data_sharing_policy.html

REFERENCES:
- [Background] Hyman DM, Piha-Paul SA, Won H, Rodon J, Saura C, Shapiro GI, Juric D, Quinn DI, Moreno V, Doger B, Mayer IA, Boni V, Calvo E, Loi S, Lockhart AC, Erinjeri JP, Scaltriti M, Ulaner GA, Patel J, Tang J, Beer H, Selcuklu SD, Hanrahan AJ, Bouvier N, Melcer M, Murali R, Schram AM, Smyth LM, Jhaveri K, Li BT, Drilon A, Harding JJ, Iyer G, Taylor BS, Berger MF, Cutler RE Jr, Xu F, Butturini A, Eli LD, Mann G, Farrell C, Lalani AS, Bryce RP, Arteaga CL, Meric-Bernstam F, Baselga J, Solit DB. HER kinase inhibition in patients with HER2- and HER3-mutant cancers. Nature. 2018 Feb 8;554(7691):189-194. doi: 10.1038/nature25475. Epub 2018 Jan 31. PMID 29420467
- [Background] Smyth LM, Piha-Paul SA, Won HH, Schram AM, Saura C, Loi S, Lu J, Shapiro GI, Juric D, Mayer IA, Arteaga CL, de la Fuente MI, Brufksy AM, Spanggaard I, Mau-Sorensen M, Arnedos M, Moreno V, Boni V, Sohn J, Schwartzberg LS, Gonzalez-Farre X, Cervantes A, Bidard FC, Gorelick AN, Lanman RB, Nagy RJ, Ulaner GA, Chandarlapaty S, Jhaveri K, Gavrila EI, Zimel C, Selcuklu SD, Melcer M, Samoila A, Cai Y, Scaltriti M, Mann G, Xu F, Eli LD, Dujka M, Lalani AS, Bryce R, Baselga J, Taylor BS, Solit DB, Meric-Bernstam F, Hyman DM. Efficacy and Determinants of Response to HER Kinase Inhibition in HER2-Mutant Metastatic Breast Cancer. Cancer Discov. 2020 Feb;10(2):198-213. doi: 10.1158/2159-8290.CD-19-0966. Epub 2019 Dec 5. PMID 31806627
- [Derived] Li BT, Gandhi L, Ravichandran V, Besse B, Mazieres J, Shapiro GI, Boni V, Waqar SN, Park H, Quinn DI, Martinez A, Stemmer SM, Cortot AB, Barlesi F, Quoix E, Burkard ME, Selcuklu SD, Hunt C, Donoghue MTA, Kris MG, Bebchuk J, Eli LD, McCulloch L, Solit DB, Janne PA. Efficacy of Neratinib-Based Therapy in ERBB2-Mutant Lung Adenocarcinomas: Findings From 2 International Phase 2 Studies. Clin Lung Cancer. 2025 Oct 1:S1525-7304(25)00234-7. doi: 10.1016/j.cllc.2025.09.009. Online ahead of print. PMID 41193346
- [Derived] Friedman CF, D'Souza A, Bello Roufai D, Tinker AV, de Miguel M, Gambardella V, Goldman J, Loi S, Melisko ME, Oaknin A, Spanggaard I, Shapiro GI, ElNaggar AC, Panni S, Ravichandran V, Frazier AL, DiPrimeo D, Eli LD, Solit DB. Targeting HER2-mutant metastatic cervical cancer with neratinib: Final results from the phase 2 SUMMIT basket trial. Gynecol Oncol. 2024 Feb;181:162-169. doi: 10.1016/j.ygyno.2023.12.004. Epub 2024 Jan 11. PMID 38211393
- [Derived] Jhaveri K, Eli LD, Wildiers H, Hurvitz SA, Guerrero-Zotano A, Unni N, Brufsky A, Park H, Waisman J, Yang ES, Spanggaard I, Reid S, Burkard ME, Vinayak S, Prat A, Arnedos M, Bidard FC, Loi S, Crown J, Bhave M, Piha-Paul SA, Suga JM, Chia S, Saura C, Garcia-Saenz JA, Gambardella V, de Miguel MJ, Gal-Yam EN, Rapael A, Stemmer SM, Ma C, Hanker AB, Ye D, Goldman JW, Bose R, Peterson L, Bell JSK, Frazier A, DiPrimeo D, Wong A, Arteaga CL, Solit DB. Neratinib + fulvestrant + trastuzumab for HR-positive, HER2-negative, HER2-mutant metastatic breast cancer: outcomes and biomarker analysis from the SUMMIT trial. Ann Oncol. 2023 Oct;34(10):885-898. doi: 10.1016/j.annonc.2023.08.003. Epub 2023 Aug 18. PMID 37597578
- [Derived] Harding JJ, Piha-Paul SA, Shah RH, Murphy JJ, Cleary JM, Shapiro GI, Quinn DI, Brana I, Moreno V, Borad M, Loi S, Spanggaard I, Park H, Ford JM, Arnedos M, Stemmer SM, de la Fouchardiere C, Fountzilas C, Zhang J, DiPrimeo D, Savin C, Duygu Selcuklu S, Berger MF, Eli LD, Meric-Bernstam F, Jhaveri K, Solit DB, Abou-Alfa GK. Antitumour activity of neratinib in patients with HER2-mutant advanced biliary tract cancers. Nat Commun. 2023 Feb 6;14(1):630. doi: 10.1038/s41467-023-36399-y. PMID 36746967
- [Derived] Shishido SN, Masson R, Xu L, Welter L, Prabakar RK, D' Souza A, Spicer D, Kang I, Jayachandran P, Hicks J, Lu J, Kuhn P. Disease characterization in liquid biopsy from HER2-mutated, non-amplified metastatic breast cancer patients treated with neratinib. NPJ Breast Cancer. 2022 Feb 18;8(1):22. doi: 10.1038/s41523-022-00390-5. PMID 35181666
- [Derived] Oaknin A, Friedman CF, Roman LD, D'Souza A, Brana I, Bidard FC, Goldman J, Alvarez EA, Boni V, ElNaggar AC, Passalacqua R, Do KTM, Santin AD, Keyvanjah K, Xu F, Eli LD, Lalani AS, Bryce RP, Hyman DM, Meric-Bernstam F, Solit DB, Monk BJ. Neratinib in patients with HER2-mutant, metastatic cervical cancer: Findings from the phase 2 SUMMIT basket trial. Gynecol Oncol. 2020 Oct;159(1):150-156. doi: 10.1016/j.ygyno.2020.07.025. Epub 2020 Jul 25. PMID 32723675
- [Derived] Ulaner GA, Saura C, Piha-Paul SA, Mayer I, Quinn D, Jhaveri K, Stone B, Shahin S, Mann G, Dujka M, Bryce R, Meric-Bernstam F, Solit DB, Hyman DM. Impact of FDG PET Imaging for Expanding Patient Eligibility and Measuring Treatment Response in a Genome-Driven Basket Trial of the Pan-HER Kinase Inhibitor, Neratinib. Clin Cancer Res. 2019 Dec 15;25(24):7381-7387. doi: 10.1158/1078-0432.CCR-19-1658. Epub 2019 Sep 23. PMID 31548342
- [Derived] Hanker AB, Brewer MR, Sheehan JH, Koch JP, Sliwoski GR, Nagy R, Lanman R, Berger MF, Hyman DM, Solit DB, He J, Miller V, Cutler RE Jr, Lalani AS, Cross D, Lovly CM, Meiler J, Arteaga CL. An Acquired HER2T798I Gatekeeper Mutation Induces Resistance to Neratinib in a Patient with HER2 Mutant-Driven Breast Cancer. Cancer Discov. 2017 Jun;7(6):575-585. doi: 10.1158/2159-8290.CD-16-1431. Epub 2017 Mar 8. PMID 28274957
- See also: HER Kinase Inhibition in Patients With HER2- And HER3-mutant Cancers — https://www.ncbi.nlm.nih.gov/pubmed/29420467
- See also: Efficacy and Determinants of Response to HER Kinase Inhibition in HER2 -Mutant Metastatic Breast Cancer — https://www.ncbi.nlm.nih.gov/pubmed/31806627

RESULTS

PARTICIPANT FLOW:
Groups:
- Neratinib: Neratinib Monotherapy (Neratinib 240 mg PO daily)
- Neratinib + Fulvestrant: Neratinib + Fulvestrant (Neratinib 240 mg PO daily + Fulvestrant 500 mg IM on Days 1, 15 of the first month, then Day 1 of every 4-week cycle)
- Neratinib + Paclitaxel: Neratinib + Paclitaxel (Neratinib 240 mg PO daily + Paclitaxel 80 mg/m2 IV on Days 1, 8, and 15 of every 4-week cycle)
- Neratinib + Trastuzumab: Neratinib + Trastuzumab (Neratinib 240 mg PO daily + Trastuzumab 8 mg/kg IV followed by 6 mg/kg IV every 3 weeks)
- Neratinib + Fulvestrant + Trastuzumab: Neratinib + Fulvestrant + Trastuzumab (Neratinib 240 mg PO daily + Fulvestrant 500 mg IM on Study Day 1, 15, and 29; once every 28 days thereafter + Trastuzumab 8 mg/kg IV followed by 6 mg/kg IV every 3 weeks)
- Fulvestrant: Fulvestrant (Fulvestrant 500 mg IM on Study Day 1, 15, and 29; once every 28 days thereafter)
- Fulvestrant + Trastuzumab: Fulvestrant + Trastuzumab (Fulvestrant 500 mg IM on Study Day 1, 15, and 29; once every 28 days thereafter + Trastuzumab 8 mg/kg IV followed by 6 mg/kg IV every 3 weeks)
Period: Overall Study
Arm/Group | Neratinib | Neratinib + Fulvestrant | Neratinib + Paclitaxel | Neratinib + Trastuzumab | Neratinib + Fulvestrant + Trastuzumab | Fulvestrant | Fulvestrant + Trastuzumab
Started | 318 | 45 | 23 | 92 | 90 | 7 | 7
Treated | 317 | 45 | 22 | 92 | 90 | 7 | 7
Completed | 231 | 31 | 14 | 70 | 32 | 2 | 0
Not Completed | 87 | 14 | 9 | 22 | 58 | 5 | 7
Not completed — Withdrawal by Subject | 23 | 3 | 3 | 5 | 6 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 18 | 3 | 0 | 5 | 3 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other, Disease progression | 2 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Discontinuation of study by sponsor | 41 | 7 | 5 | 12 | 46 | 5 | 6
Not completed — Not Treated | 1 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neratinib | Neratinib + Fulvestrant | Neratinib + Paclitaxel | Neratinib + Trastuzumab | Neratinib + Fulvestrant + Trastuzumab | Fulvestrant | Fulvestrant + Trastuzumab | Total
Number analyzed (Participants) | 317 | 45 | 22 | 92 | 90 | 7 | 7 | 580
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 201 | 28 | 4 | 57 | 59 | 6 | 3 | 358
  >=65 years | 116 | 17 | 18 | 35 | 31 | 1 | 4 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (13.1) | 60.6 (11.5) | 69.4 (9.4) | 60.4 (11.1) | 59.2 (11.6) | 58.3 (11.2) | 62.0 (12.4) | 60.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 188 | 45 | 5 | 58 | 89 | 7 | 7 | 399
  Male | 129 | 0 | 17 | 34 | 1 | 0 | 0 | 181
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 255 | 38 | 21 | 70 | 77 | 7 | 5 | 473
  Race: Asian | 18 | 2 | 0 | 7 | 1 | 0 | 0 | 28
  Race: Black or African American | 16 | 1 | 0 | 4 | 4 | 0 | 1 | 26
  Race: American Indian or Alaska Native | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 3
  Race: Other | 6 | 1 | 0 | 2 | 0 | 0 | 0 | 9
  Race: Unknown | 7 | 1 | 0 | 4 | 1 | 0 | 0 | 13
  Race: Not Reported | 13 | 2 | 1 | 5 | 7 | 0 | 0 | 28
Tumor type [Count of Participants; unit: Participants] — Cohort by tumor type
  Participants
    Breast cancer HR+ or HR- | 36 | 0 | 0 | 0 | 0 | 0 | 0 | 36
    Breast cancer HR+ | 0 | 45 | 0 | 0 | 31 | 0 | 0 | 76
    Breast cancer HR+, prior CDK46 inhibitors | 0 | 0 | 0 | 0 | 59 | 7 | 7 | 73
    Breast cancer HR- | 0 | 0 | 0 | 21 | 0 | 0 | 0 | 21
    Lung Her2 mutant cancer | 26 | 0 | 0 | 52 | 0 | 0 | 0 | 78
    Lung EGFR mutant exon 18 cancer | 31 | 0 | 0 | 0 | 0 | 0 | 0 | 31
    Biliary tract cancer | 25 | 0 | 0 | 0 | 0 | 0 | 0 | 25
    Cervical cancer | 22 | 0 | 0 | 0 | 0 | 0 | 0 | 22
    Bladder/Urinary Tract cancer | 16 | 0 | 22 | 0 | 0 | 0 | 0 | 38
    Brain EGFR mutant cancer | 38 | 0 | 0 | 0 | 0 | 0 | 0 | 38
    Colorectal cancer | 12 | 0 | 0 | 19 | 0 | 0 | 0 | 31
    Salivary gland cancer | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 11
    Endometrial cancer | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 7
    Fibrolamellar carcinoma (FLC) | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 15
    Gastroesophageal cancer | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 7
    Ovarian cancer | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 10
    HER2 NOS cancer | 42 | 0 | 0 | 0 | 0 | 0 | 0 | 42
    HER3 NOS cancer | 16 | 0 | 0 | 0 | 0 | 0 | 0 | 16
    HER4 NOS cancer | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response Rate (ORR) by Independent Central Review (Breast Cancer With Prior CDK46i Cohort)
Description: Percentage of participants who are confirmed by independent central review to have achieved complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 (HR+, HER2 negative metastatic breast cancer cohorts).
  Per Response Evaluation Criteria in Sold Tumors Criteria (RECISTv1.1) for target lesions and assessed by MRI or CT: Complete response(CR),Disappearance of all target lesions; Partial response(PR),>=30% decrease in sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: From enrollment date to first confirmed Complete or Partial Response, whichever came earlier, assessed up to 58 months
Population: Cohort of cancer type and treatment
Measure: Number; unit: percentage of participants
Groups:
- Breast HR+ w Prior CDK4/6i (Neratinib + Fulvestrant + Trastuzumab): Consisting of 33 patients from the randomized cohort and 26 from the non-randomized cohort in breast cancer who had prior CDK4/6 inhibitor, treated with (Neratinib + Fulvestrant + Trastuzumab)
- Breast HR+ w. Prior CDK4/6i (Fulvestrant): Breast HR+ with Prior CDK4/6 inhibitor patients treated with Fulvestrant Monotherapy
- Breast HR+ With Prior CDK4/6i (Fulvestrant + Trastuzumab): Breast cancer HR+ w prior CDK4/6 inhibitor patients treated with combination of (Fulvestrant + Trastuzumab)
Arm/Group | Breast HR+ w Prior CDK4/6i (Neratinib + Fulvestrant + Trastuzumab) | Breast HR+ w. Prior CDK4/6i (Fulvestrant) | Breast HR+ With Prior CDK4/6i (Fulvestrant + Trastuzumab)
Number analyzed (Participants) | 59 | 7 | 7
percentage of participants | 40.7 | 0 | 14.3

2. Primary Outcome: Confirmed Objective Response Rate (ORR) by Investigator Review (Cervical Cancer Cohort)
Description: Percentage of participants who are confirmed by investigator review to have achieved complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 (cervical cancer cohort).
  Per Response Evaluation Criteria in Sold Tumors Criteria (RECISTv1.1) for target lesions and assessed by MRI or CT: Complete response(CR),Disappearance of all target lesions; Partial response(PR),>=30% decrease in sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: From enrollment date to first confirmed Complete or Partial Response, whichever came earlier, assessed up to 58 months
Population: Cohort of cancer type and treatment
Measure: Number; unit: percentage of participants
Groups:
- Cervical (Neratinib): Cervical cancer patients treated with Neratinib Monotherapy
Arm/Group | Cervical (Neratinib)
Number analyzed (Participants) | 22
percentage of participants | 18.2

3. Primary Outcome: Objective Response Rate (ORR) at First Assessment by Investigator Review (All Other Cohorts)
Description: Percentage of participants who achieve CR or PR per Response Evaluation Criteria in Sold Tumors Criteria (RECIST) v1.1, or other defined response criteria, at the first scheduled tumor assessment (all other cohorts), per RECIST (if assessed) or PERCIST.
  RECISTv1.1 for target lesions and assessed by MRI or CT: Complete response(CR),Disappearance of all target lesions; Partial response(PR),>=30% decrease in sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
  PERCISTv1.0: Complete Metabolic Response - Complete resolution of 18F-FDG uptake within measurable target lesion so that it is less than mean liver activity and indistinguishable from surrounding background blood-pool levels
  Partial Metabolic Response - Reduction of minimum of 30% in target measurable tumour 18F-FDG SULpeak. Absolute drop in SUL must be at least 0.8 SUL units, as well. No new lesions.
  Positive Metabolic Response - Participants having either "Complete Metabolic Response" or "Part
Time Frame: From first treatment date to first Complete or Partial Response, whichever came earlier, assessed up to 8 or 9 weeks
Population: Cohort of cancer type and treatment
Measure: Number; unit: percentage of participant
Groups:
- Breast Cancer (Neratinib): Breast cancer HR+ or HR- patients treated with Neratinib Monotherapy
- Breast Cancer HR+ (Neratinib + Fulvestrant): Breast cancer HR+ patients treated with combination of (Neratinib + Fulvestrant)
- Breast Cancer HR+ (Neratinib + Fulvestrant + Trastuzumab): Breast cancer HR+ patients treated with combination of (Neratinib + Fulvestrant + Trastuzumab)
- Breast Cancer HR- (Neratinib + Trastuzumab): Breast cancer HR- patients treated with combination of (Neratinib + Trastuzumab)
- Lung Cancer HER2 Mutant (Neratinib): NSCLC Lung cancer HER2 mutant patients treated with Neratinib Monotherapy
- Lung Cancer HER2 Mutant (Neratinib + Trastuzumab): NSCLC Lung cancer HER2 mutant patients treated with combination of (Neratinib + Trastuzumab)
- Lung Cancer EGFR Mutant Exon 18 (Neratinib): NSCLC Lung cancer EGFR mutant exon 18 patients treated with Neratinib Monotherapy
- Biliary Tract Cancer (Neratinib): Biliary tract cancer patients treated with Neratinib Monotherapy
- Bladder/Urinary Tract Cancer (Neratinib): Bladder/Urinary Tract cancer patients treated with Neratinib Monotherapy
- Bladder/Urinary Tract Cancer (Neratinib + Paclitaxel): Bladder/Urinary Tract cancer patients treated with combination of (Neratinib + Paclitaxel)
- Brain Cancer (Neratinib): Primary brain tumors (glioblastoma multiforme (GBM), gliosarcoma, and/or Grade III glioma) patients treated with Neratinib Monotherapy
- Colorectal Cancer (Neratinib): Colorectal cancer patients treated with Neratinib Monotherapy
- Colorectal Cancer (Neratinib + Trastuzumab): Colorectal cancer patients treated with combination of (Neratinib + Trastuzumab)
- Endometrial Cancer (Neratinib): Endometrial cancer patients treated with Neratinib Monotherapy
- Ovarian Cancer (Neratinib): Ovarian cancer patients treated with Neratinib Monotherapy
- Salivary Gland Cancer (Neratinib): Salivary gland cancer patients treated with Neratinib Monotherapy
- Gastroesophageal Cancer (Neratinib): Gastroesophageal cancer patients treated with Neratinib Monotherapy
- Fibrolamellar Carcinoma (FLC) (Neratinib): Fibrolamellar carcinoma (FLC) patients treated with Neratinib Monotherapy
- HER2 NOS Cancer (Neratinib): HER2 mutant Solid tumors, not otherwise specified (NOS) patients treated with Neratinib Monotherapy
- HER3 NOS Cancer (Neratinib): HER3 mutant Solid tumors, not otherwise specified (NOS) patients treated with Neratinib Monotherapy
- HER4 NOS Cancer (Neratinib): HER4 mutant Solid tumors, not otherwise specified (NOS) patients treated with Neratinib Monotherapy
Arm/Group | Breast Cancer (Neratinib) | Breast Cancer HR+ (Neratinib + Fulvestrant) | Breast Cancer HR+ (Neratinib + Fulvestrant + Trastuzumab) | Breast Cancer HR- (Neratinib + Trastuzumab) | Lung Cancer HER2 Mutant (Neratinib) | Lung Cancer HER2 Mutant (Neratinib + Trastuzumab) | Lung Cancer EGFR Mutant Exon 18 (Neratinib) | Biliary Tract Cancer (Neratinib) | Bladder/Urinary Tract Cancer (Neratinib) | Bladder/Urinary Tract Cancer (Neratinib + Paclitaxel) | Brain Cancer (Neratinib) | Colorectal Cancer (Neratinib) | Colorectal Cancer (Neratinib + Trastuzumab) | Endometrial Cancer (Neratinib) | Ovarian Cancer (Neratinib) | Salivary Gland Cancer (Neratinib) | Gastroesophageal Cancer (Neratinib) | Fibrolamellar Carcinoma (FLC) (Neratinib) | HER2 NOS Cancer (Neratinib) | HER3 NOS Cancer (Neratinib) | HER4 NOS Cancer (Neratinib)
Number analyzed (Participants) | 36 | 45 | 31 | 21 | 26 | 52 | 31 | 25 | 16 | 22 | 38 | 12 | 19 | 7 | 10 | 11 | 7 | 15 | 42 | 16 | 3
percentage of participant | 36.1 | 42.2 | 48.4 | 33.3 | 3.8 | 15.4 | 19.4 | 12.0 | 0 | 13.6 | 0 | 0 | 5.3 | 0 | 0 | 36.4 | 0 | 0 | 4.8 | 0 | 0

4. Secondary Outcome: Confirmed Objective Response Rate (ORR) by Investigator Review (Breast Cancer With Prior CDK46i Cohort)
Description: Percentage of participants who are confirmed by investigator review to have achieved complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 (HR+, HER2 negative metastatic breast cancer cohorts).
  Per Response Evaluation Criteria in Sold Tumors Criteria (RECISTv1.1) for target lesions and assessed by MRI or CT: Complete response(CR),Disappearance of all target lesions; Partial response(PR),>=30% decrease in sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: From enrollment date to first confirmed Complete or Partial Response, whichever came earlier, assessed up to 58 months
Population: Cohort of cancer type and treatment
Measure: Number; unit: percentage of participants
Arm/Group | Breast HR+ w Prior CDK4/6i (Neratinib + Fulvestrant + Trastuzumab) | Breast HR+ w. Prior CDK4/6i (Fulvestrant) | Breast HR+ With Prior CDK4/6i (Fulvestrant + Trastuzumab)
Number analyzed (Participants) | 59 | 7 | 7
percentage of participants | 30.5 | 0 | 0

5. Secondary Outcome: Confirmed Objective Response Rate (ORR) by Investigator Review (All Other Cohorts)
Description: Percentage of participants who achieve CR or PR per RECIST v1.1, or metabolic complete response via PERCIST v1.0.
  For RECIST, A complete or partial response that is confirmed no less than 4-weeks after the criteria for response are initially met. PERCIST criteria were used for patients without RECIST assessments.
Time Frame: From first treatment date to confirmed Complete or Partial Response, assessed up to 58 months.
Measure: Number; unit: percentage of participant
Arm/Group | Breast Cancer (Neratinib) | Breast Cancer HR+ (Neratinib + Fulvestrant) | Breast Cancer HR+ (Neratinib + Fulvestrant + Trastuzumab) | Breast Cancer HR- (Neratinib + Trastuzumab) | Lung Cancer HER2 Mutant (Neratinib) | Lung Cancer HER2 Mutant (Neratinib + Trastuzumab) | Lung Cancer EGFR Mutant Exon 18 (Neratinib) | Biliary Tract Cancer (Neratinib) | Bladder/Urinary Tract Cancer (Neratinib) | Bladder/Urinary Tract Cancer (Neratinib + Paclitaxel) | Brain Cancer (Neratinib) | Colorectal Cancer (Neratinib) | Colorectal Cancer (Neratinib + Trastuzumab) | Endometrial Cancer (Neratinib) | Ovarian Cancer (Neratinib) | Salivary Gland Cancer (Neratinib) | Gastroesophageal Cancer (Neratinib) | Fibrolamellar Carcinoma (FLC) (Neratinib) | HER2 NOS Cancer (Neratinib) | HER3 NOS Cancer (Neratinib) | HER4 NOS Cancer (Neratinib)
Number analyzed (Participants) | 36 | 45 | 31 | 21 | 26 | 52 | 31 | 25 | 16 | 22 | 38 | 12 | 19 | 7 | 10 | 11 | 7 | 15 | 42 | 16 | 3
percentage of participant | 25.0 | 28.9 | 35.5 | 33.3 | 3.8 | 9.6 | 32.3 | 16.0 | 0 | 13.6 | 2.6 | 0 | 5.3 | 0 | 0 | 9.1 | 0 | 0 | 2.4 | 0 | 0

6. Secondary Outcome: Duration of Response (DOR) by Independent Central Review (Breast Cancer With Prior CDK46i Cohort)
Description: Time from which measurement criteria are met for response (whichever status is recorded first) until the first date of documented disease progression or death. Disease progression assessed by RECIST criteria, or for PERCIST for those participants who did not have RECIST performed.
Time Frame: From first response to first disease progression or death, assessed up to 58 months
Population: Number of confirmed responders
Measure: Median (95% Confidence Interval); unit: month
Groups:
- Breast Cancer HR+ w Prior CDK4/6i (Neratinib + Fulvestrant + Trastuzumab): Breast cancer HR+ patients having prior CDK4/6i treated with combination of (Neratinib + Fulvestrant + Trastuzumab)
- Breast Cancer HR+ w Prior CDK4/6i (Fulvestrant): Breast cancer HR+ patients having prior CDK4/6i treated with Fulvestrant Monotherapy
- Breast Cancer HR+ w Prior CDK4/6i (Fulvestrant + Trastuzumab): Breast cancer HR+ patients having prior CDK4/6i treated with combination of (Fulvestrant + Trastuzumab)
Arm/Group | Breast Cancer HR+ w Prior CDK4/6i (Neratinib + Fulvestrant + Trastuzumab) | Breast Cancer HR+ w Prior CDK4/6i (Fulvestrant) | Breast Cancer HR+ w Prior CDK4/6i (Fulvestrant + Trastuzumab)
Number analyzed (Participants) | 24 | 0 | 1
month | 13.14 [6.41 to NA] — Upper limits of 95% Confidence Interval (CI) was not estimable due to insufficient number of events. |  | NA [NA to NA] — Median and Upper, lower limits of 95% Confidence Interval (CI) were not estimable due to insufficient number of events.

7. Secondary Outcome: Duration of Response (DOR) by Investigator Review (All Cohorts)
Description: as for outcome 6
Time Frame: From first response to first disease progression or death, assessed up to 58 months
Population: Number of confirmed responders
Measure: Median (95% Confidence Interval); unit: month
Groups:
- Cervical Cancer (Neratinib): Cervical cancer patients treated with Neratinib Monotherapy
Arm/Group | Breast Cancer HR+ w Prior CDK4/6i (Neratinib + Fulvestrant + Trastuzumab) | Breast Cancer HR+ w Prior CDK4/6i (Fulvestrant) | Breast Cancer HR+ w Prior CDK4/6i (Fulvestrant + Trastuzumab) | Breast Cancer (Neratinib) | Breast Cancer HR+ (Neratinib + Fulvestrant) | Breast Cancer HR+ (Neratinib + Fulvestrant + Trastuzumab) | Breast Cancer HR- (Neratinib + Trastuzumab) | Cervical Cancer (Neratinib) | Lung Cancer HER2 Mutant (Neratinib) | Lung Cancer HER2 Mutant (Neratinib + Trastuzumab) | Lung Cancer EGFR Mutant Exon 18 (Neratinib) | Biliary Tract Cancer (Neratinib) | Bladder/Urinary Tract Cancer (Neratinib) | Bladder/Urinary Tract Cancer (Neratinib + Paclitaxel) | Brain Cancer (Neratinib) | Colorectal Cancer (Neratinib) | Colorectal Cancer (Neratinib + Trastuzumab) | Endometrial Cancer (Neratinib) | Ovarian Cancer (Neratinib) | Salivary Gland Cancer (Neratinib) | Gastroesophageal Cancer (Neratinib) | Fibrolamellar Carcinoma (FLC) (Neratinib) | HER2 NOS Cancer (Neratinib) | HER3 NOS Cancer (Neratinib) | HER4 NOS Cancer (Neratinib)
Number analyzed (Participants) | 23 | 0 | 0 | 9 | 13 | 11 | 7 | 4 | 1 | 5 | 10 | 4 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
month | 14.4 [7.8 to 18.6] |  |  | 4.76 [3.71 to 16.62] | 9.23 [5.49 to 38.97] | 9.17 [4.14 to NA] — Upper limits of 95% Confidence Interval (CI) was not estimable due to insufficient number of events. | 7.28 [4.17 to NA] — Upper limits of 95% Confidence Interval (CI) was not estimable due to insufficient number of events. | 7.62 [5.55 to 12.25] | 9.23 [NA to NA] — Upper and lower limits of 95% Confidence Interval (CI) were not estimable due to insufficient number of events. | 6.80 [4.17 to NA] — Upper limits of 95% Confidence Interval (CI) was not estimable due to insufficient number of events. | 22.24 [4.01 to 30.03] | 3.75 [2.99 to 4.67] |  | 7.20 [2.76 to 7.59] | 19.94 [NA to NA] — Upper and lower limits of 95% Confidence Interval (CI) were not estimable due to insufficient number of events. |  | 12.19 [NA to NA] — Upper and lower limits of 95% Confidence Interval (CI) were not estimable due to insufficient number of events. |  |  | NA [NA to NA] — Median and Upper, lower limits of 95% Confidence Interval (CI) were not estimable due to insufficient number of events. |  |  | 3.71 [NA to NA] — Upper and lower limits of 95% Confidence Interval (CI) were not estimable due to insufficient number of events. |  |

8. Secondary Outcome: Clinical Benefit Rate (CBR) by Independent Central Review (Breast Cancer With Prior CDK46i Cohort)
Description: Percentage of participants with CR + PR + stable disease ≥16, or ≥24 weeks for breast cancer, from the date of enrollment.
Time Frame: From enrollment date to first documented response or stable disease ≥16, or ≥24 weeks for breast cancer, assessed up to 58 months
Measure: Number; unit: percentage of participant
Arm/Group | Breast Cancer HR+ w Prior CDK4/6i (Neratinib + Fulvestrant + Trastuzumab) | Breast Cancer HR+ w Prior CDK4/6i (Fulvestrant) | Breast Cancer HR+ w Prior CDK4/6i (Fulvestrant + Trastuzumab)
Number analyzed (Participants) | 59 | 7 | 7
percentage of participant | 49.2 | 0 | 14.3

9. Secondary Outcome: Clinical Benefit Rate (CBR) by Investigator Review (All Cohorts)
Description: as for outcome 8
Time Frame: as for outcome 8
Measure: Number; unit: percentage of participant
Arm/Group | Breast Cancer HR+ w Prior CDK4/6i (Neratinib + Fulvestrant + Trastuzumab) | Breast Cancer HR+ w Prior CDK4/6i (Fulvestrant) | Breast Cancer HR+ w Prior CDK4/6i (Fulvestrant + Trastuzumab) | Breast Cancer (Neratinib) | Breast Cancer HR+ (Neratinib + Fulvestrant) | Breast Cancer HR+ (Neratinib + Fulvestrant + Trastuzumab) | Breast Cancer HR- (Neratinib + Trastuzumab) | Cervical Cancer (Neratinib) | Lung Cancer HER2 Mutant (Neratinib) | Lung Cancer HER2 Mutant (Neratinib + Trastuzumab) | Lung Cancer EGFR Mutant Exon 18 (Neratinib) | Biliary Tract Cancer (Neratinib) | Bladder/Urinary Tract Cancer (Neratinib) | Bladder/Urinary Tract Cancer (Neratinib + Paclitaxel) | Brain Cancer (Neratinib) | Colorectal Cancer (Neratinib) | Colorectal Cancer (Neratinib + Trastuzumab) | Endometrial Cancer (Neratinib) | Ovarian Cancer (Neratinib) | Salivary Gland Cancer (Neratinib) | Gastroesophageal Cancer (Neratinib) | Fibrolamellar Carcinoma (FLC) (Neratinib) | HER2 NOS Cancer (Neratinib) | HER3 NOS Cancer (Neratinib) | HER4 NOS Cancer (Neratinib)
Number analyzed (Participants) | 59 | 7 | 7 | 36 | 45 | 31 | 21 | 22 | 26 | 52 | 31 | 25 | 16 | 22 | 38 | 12 | 19 | 7 | 10 | 11 | 7 | 15 | 42 | 16 | 3
percentage of participant | 54.2 | 0 | 0 | 33.3 | 42.2 | 54.8 | 42.9 | 45.5 | 38.5 | 30.8 | 48.4 | 24.0 | 18.8 | 31.8 | 10.5 | 8.3 | 21.1 | 14.3 | 20.0 | 54.5 | 0 | 13.3 | 19.0 | 6.3 | 0

10. Secondary Outcome: Progression-Free Survival (PFS) by Independent Central Review (Breast Cancer With Prior CDK46i Cohort)
Description: Number of months between first dose date and the first date on which recurrence, progression, or death due to any cause, is documented, censored at the last tumor assessment or at the initiation of new anticancer therapy. Progression was defined by RECIST criteria for those participants with RECIST assessments; and PERCIST criteria for other participants.
Time Frame: From enrollment date until the date of first documented progression, or date of death from any cause, whichever came first, assessed up to 58 months
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Breast Cancer HR+ w Prior CDK4/6i (Neratinib + Fulvestrant + Trastuzumab) | Breast Cancer HR+ w Prior CDK4/6i (Fulvestrant) | Breast Cancer HR+ w Prior CDK4/6i (Fulvestrant + Trastuzumab)
Number analyzed (Participants) | 59 | 7 | 7
month | 8.11 [6.01 to 16.39] | 2.27 [1.61 to NA] — Upper limit of 95% Confidence Interval (CI) was not estimable due to insufficient number of events. | 4.11 [1.87 to 4.11]

11. Secondary Outcome: Progression-Free Survival (PFS) by Investigator Review (All Cohorts)
Description: as for outcome 10
Time Frame: as for outcome 10
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Breast Cancer HR+ w Prior CDK4/6i (Neratinib + Fulvestrant + Trastuzumab) | Breast Cancer HR+ w Prior CDK4/6i (Fulvestrant) | Breast Cancer HR+ w Prior CDK4/6i (Fulvestrant + Trastuzumab) | Breast Cancer (Neratinib) | Breast Cancer HR+ (Neratinib + Fulvestrant) | Breast Cancer HR+ (Neratinib + Fulvestrant + Trastuzumab) | Breast Cancer HR- (Neratinib + Trastuzumab) | Cervical Cancer (Neratinib) | Lung Cancer HER2 Mutant (Neratinib) | Lung Cancer HER2 Mutant (Neratinib + Trastuzumab) | Lung Cancer EGFR Mutant Exon 18 (Neratinib) | Biliary Tract Cancer (Neratinib) | Bladder/Urinary Tract Cancer (Neratinib) | Bladder/Urinary Tract Cancer (Neratinib + Paclitaxel) | Brain Cancer (Neratinib) | Colorectal Cancer (Neratinib) | Colorectal Cancer (Neratinib + Trastuzumab) | Endometrial Cancer (Neratinib) | Ovarian Cancer (Neratinib) | Salivary Gland Cancer (Neratinib) | Gastroesophageal Cancer (Neratinib) | Fibrolamellar Carcinoma (FLC) (Neratinib) | HER2 NOS Cancer (Neratinib) | HER3 NOS Cancer (Neratinib) | HER4 NOS Cancer (Neratinib)
Number analyzed (Participants) | 59 | 7 | 7 | 36 | 45 | 31 | 21 | 22 | 26 | 52 | 31 | 25 | 16 | 22 | 38 | 12 | 19 | 7 | 10 | 11 | 7 | 15 | 42 | 16 | 3
month | 8.3 [6.0 to 12.7] | 4.1 [1.6 to 4.1] | 3.9 [1.9 to 4.1] | 3.48 [1.94 to 3.88] | 5.36 [3.71 to 9.23] | 8.21 [4.07 to 11.01] | 6.24 [2.10 to 10.25] | 5.09 [1.74 to 7.23] | 4.17 [1.87 to 8.80] | 4.01 [2.10 to 4.57] | 5.75 [2.27 to 9.23] | 2.76 [1.05 to 3.75] | 1.77 [1.68 to 3.55] | 3.75 [1.87 to 5.62] | 1.81 [1.02 to 2.69] | 1.71 [1.45 to 1.87] | 2.04 [1.81 to 3.48] | 1.87 [1.61 to 6.87] | 2.37 [1.48 to 7.36] | 5.32 [1.81 to 9.26] | 1.74 [0.82 to 2.23] | 3.58 [1.84 to 3.71] | 1.84 [1.74 to 2.07] | 1.69 [1.41 to 2.04] | 1.71 [1.12 to 1.74]

12. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: The safety of neratinib in patients as measured by the incidence of treatment-emergent adverse events (TEAE), including serious adverse events (SAEs), in study participants. TEAEs are any adverse event that occurred on or after first dose of investigational product and up to 28 days after the last dose
Time Frame: From first dose through 28 days after the last dose, assessed up to 75 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Neratinib | Neratinib + Fulvestrant | Neratinib + Paclitaxel | Neratinib + Trastuzumab | Neratinib + Fulvestrant + Trastuzumab | Fulvestrant | Fulvestrant + Trastuzumab
Number analyzed (Participants) | 317 | 45 | 22 | 92 | 90 | 7 | 7
Participants
  Any treatment-emergent adverse event | 313 | 45 | 21 | 92 | 89 | 7 | 7
  Any treatment-emergent serious adverse event | 144 | 12 | 13 | 45 | 28 | 5 | 0

ADVERSE EVENTS:
Time Frame: All events from day 1 of study drug through 28 days after last dose are included, up to 75 months.
Arm/Group | Neratinib | Neratinib + Fulvestrant | Neratinib + Paclitaxel | Neratinib + Trastuzumab | Neratinib + Fulvestrant + Trastuzumab | Fulvestrant | Fulvestrant + Trastuzumab
All-Cause Mortality (participants affected / at risk) | 231/317 | 31/45 | 14/22 | 71/92 | 32/90 | 2/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 144/317 | 12/45 | 13/22 | 45/92 | 28/90 | 5/7 | 0/7
Other Adverse Events (participants affected / at risk) | 304/317 | 45/45 | 20/22 | 92/92 | 89/90 | 7/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib (N=317) | Neratinib + Fulvestrant (N=45) | Neratinib + Paclitaxel (N=22) | Neratinib + Trastuzumab (N=92) | Neratinib + Fulvestrant + Trastuzumab (N=90) | Fulvestrant (N=7) | Fulvestrant + Trastuzumab (N=7)
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 2 | 0 | 1 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 17 | 0 | 3 | 3 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 30 | 1 | 6 | 12 | 6 | 3 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 2 | 1 | 2 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 9 | 0 | 1 | 2 | 0 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 14 | 1 | 2 | 6 | 3 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0 | 2 | 0 | 1 | 0
Fatigue (General disorders) | 3 | 0 | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 3 | 0 | 1 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 7 | 0 | 0 | 3 | 1 | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malignant biliary obstruction (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 0 | 0 | 4 | 1 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 6 | 0 | 0 | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 8 | 0 | 2 | 1 | 3 | 0 | 0
Vascular device infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 1 | 2 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 0 | 1 | 2 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 2 | 0 | 0 | 1 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 4 | 0 | 0 | 1 | 2 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 10 | 0 | 1 | 1 | 3 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2 | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Brain oedema (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0
Coma (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neurological decompensation (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Device malfunction (Product Issues) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Drug abuse (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 5 | 0 | 4 | 6 | 4 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 0 | 2 | 3 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mammoplasty (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain management (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aortic thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 3 | 0 | 0 | 2 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib (N=317) | Neratinib + Fulvestrant (N=45) | Neratinib + Paclitaxel (N=22) | Neratinib + Trastuzumab (N=92) | Neratinib + Fulvestrant + Trastuzumab (N=90) | Fulvestrant (N=7) | Fulvestrant + Trastuzumab (N=7)
Anaemia (Blood and lymphatic system disorders) | 44 | 7 | 4 | 17 | 13 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 3 | 2 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 4 | 0 | 0 | 0 | 1 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 0 | 0 | 1 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 2 | 0 | 0 | 0 | 5 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 13 | 2 | 1 | 4 | 9 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 60 | 8 | 5 | 12 | 26 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 5 | 1 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 9 | 3 | 0 | 7 | 8 | 1 | 0
Constipation (Gastrointestinal disorders) | 111 | 17 | 7 | 28 | 34 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 211 | 39 | 16 | 74 | 82 | 6 | 6
Dry mouth (Gastrointestinal disorders) | 16 | 3 | 2 | 1 | 6 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 14 | 4 | 3 | 8 | 10 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 8 | 1 | 0 | 2 | 5 | 0 | 0
Flatulence (Gastrointestinal disorders) | 4 | 0 | 0 | 1 | 4 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 | 3 | 2 | 2 | 5 | 0 | 0
Nausea (Gastrointestinal disorders) | 133 | 19 | 11 | 43 | 59 | 3 | 3
Stomatitis (Gastrointestinal disorders) | 16 | 4 | 0 | 12 | 13 | 1 | 0
Vomiting (Gastrointestinal disorders) | 105 | 10 | 10 | 42 | 44 | 1 | 2
Asthenia (General disorders) | 26 | 4 | 4 | 11 | 17 | 1 | 0
Chills (General disorders) | 10 | 0 | 2 | 5 | 9 | 1 | 1
Fatigue (General disorders) | 98 | 12 | 10 | 33 | 33 | 2 | 1
Induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 21 | 8 | 1 | 8 | 10 | 0 | 0
Pain (General disorders) | 10 | 1 | 2 | 1 | 5 | 1 | 0
Pyrexia (General disorders) | 27 | 5 | 3 | 15 | 7 | 1 | 1
Food allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0 | 0 | 1 | 7 | 0 | 0
Paronychia (Infections and infestations) | 7 | 4 | 0 | 7 | 8 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 5 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 21 | 3 | 3 | 5 | 12 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2 | 5 | 0 | 0
Alanine aminotransferase increased (Investigations) | 27 | 2 | 1 | 6 | 5 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 31 | 4 | 2 | 4 | 8 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 19 | 0 | 2 | 4 | 4 | 0 | 0
Blood creatinine increased (Investigations) | 14 | 1 | 6 | 6 | 9 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 0 | 1 | 6 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1 | 1 | 2 | 1 | 0
Lymphocyte count decreased (Investigations) | 7 | 1 | 1 | 3 | 2 | 0 | 1
Neutrophil count decreased (Investigations) | 5 | 1 | 2 | 2 | 2 | 0 | 0
Weight decreased (Investigations) | 34 | 5 | 1 | 15 | 14 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 84 | 13 | 6 | 25 | 34 | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 20 | 2 | 4 | 3 | 7 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 2 | 0 | 5 | 3 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 8 | 1 | 2 | 1 | 2 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 | 1 | 1 | 6 | 4 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 4 | 1 | 5 | 5 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 15 | 1 | 1 | 7 | 12 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 11 | 3 | 0 | 5 | 7 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 9 | 2 | 2 | 4 | 4 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 11 | 0 | 1 | 2 | 7 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 7 | 5 | 12 | 11 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 28 | 8 | 3 | 11 | 7 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 2 | 4 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 4 | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 | 3 | 0 | 5 | 15 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 8 | 1 | 2 | 2 | 5 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 12 | 3 | 1 | 3 | 4 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 2 | 4 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 5 | 2 | 2 | 12 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 6 | 0 | 8 | 6 | 1 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 21 | 4 | 4 | 9 | 6 | 1 | 0
Dysgeusia (Nervous system disorders) | 18 | 2 | 4 | 5 | 9 | 0 | 1
Dysmetria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 30 | 8 | 0 | 6 | 17 | 2 | 1
Neuropathy peripheral (Nervous system disorders) | 5 | 0 | 5 | 0 | 4 | 0 | 0
Paraesthesia (Nervous system disorders) | 4 | 3 | 1 | 1 | 5 | 1 | 0
Anxiety (Psychiatric disorders) | 13 | 0 | 1 | 4 | 4 | 1 | 0
Daydreaming (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 7 | 1 | 2 | 2 | 5 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 12 | 6 | 3 | 5 | 5 | 1 | 0
Mood swings (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 3 | 2 | 2 | 0 | 3 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 4 | 2 | 10 | 8 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 | 7 | 3 | 12 | 8 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 1 | 2 | 6 | 6 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 0 | 2 | 4 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 3 | 2 | 3 | 4 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 11 | 1 | 3 | 11 | 5 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 20 | 8 | 1 | 4 | 9 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 1 | 4 | 0 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 2 | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 2 | 6 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 18 | 4 | 1 | 3 | 8 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 26 | 7 | 4 | 12 | 13 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11 | 5 | 0 | 4 | 6 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 4 | 5 | 0 | 0 | 8 | 1 | 0
Hypertension (Vascular disorders) | 19 | 3 | 1 | 8 | 10 | 0 | 2
Lymphoedema (Vascular disorders) | 3 | 3 | 0 | 2 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/26/NCT01953926/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/26/NCT01953926/SAP_001.pdf
  • Informed Consent Form: Breast (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT01953926/ICF_002.pdf
  • Informed Consent Form: Neratinib Monotherapy (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT01953926/ICF_003.pdf